CLINICAL TRIAL: NCT00614835
Title: A Pilot Study of Adjuvant Docetaxel Plus Gemcitabine in Patients With Completely Resected Leiomyosarcoma (LMS) of the Uterus
Brief Title: Adjuvant Docetaxel Plus Gemcitabine in Patients With Completely Resected Leiomyosarcoma (LMS) of the Uterus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-098
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Uterine Leiomyosarcoma; Uterine Cancer
Keywords: Gemcitabine; Docetaxel; uterine sarcoma
MeSH Terms: conditions — Uterine Neoplasms | interventions — Docetaxel; Gemcitabine

ARMS (1):
- 1 patients with completely resected uterine leiomyosarcoma (Experimental): Docetaxel plus Gemcitabine
  Interventions: Drug: Docetaxel plus Gemcitabine

INTERVENTIONS:
Drug: Docetaxel plus Gemcitabine — Gemcitabine 900 mg/m2 IV over 90 minutes day 1 Gemcitabine 900 mg/m2 IV over 90 minutes day 8 + Docetaxel 75 mg/m2 IVPB day 8 Dexamethasone 8 mg po bid days 7-9 GCSF 150 ug/m2 (round to nearest vial size: 350 ug or 480 ug) SQ days 9-15 Repeat every 21 days for total of 4 cycles

SUMMARY:
This is a pilot study of adjuvant therapy for patients with leiomyosarcoma of the uterus that has been completely removed by surgery. "Adjuvant" therapy means that the tumor (the leiomyosarcoma) has been completely removed by surgery; thus, giving further treatment now is done in hopes of decreasing the chance that the tumor will come back (relapse or recur). The main goal of this study is to show that this series of treatments is safe for patients with your type of tumor.

In this trial you will be getting drugs that have been approved for use in some types of cancer. In this study we wish to see whether the combination of two chemotherapy drugs, docetaxel and gemcitabine can decrease the chance of your tumor, leiomyosarcoma of the uterus, from coming back (relapsing). We will also be looking at the short-term side effects and risks of the drugs given in this combination to patients with leiomyosarcoma that has been completely resected (removed by surgery).

The combination of gemcitabine and docetaxel has been shown to be safe, and it has been shown to decrease the size of leiomyosarcoma tumors in patients with leiomyosarcoma of the uterus that has relapsed, or has continued to grow despite treatment with other chemotherapy drugs.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed leiomyosarcoma of the uterus, completely resected, stage I, II, III or IV within 8 weeks of surgery to remove the tumor(s). Patients with stage I tumors should have LMS that is considered high-grade by histology.
* No prior chemotherapy for LMS
* No prior treatment with gemcitabine or docetaxel Age > 18 years
* Karnofsky performance status (KPS) > or equal to 80%
* Pre-treatment absolute neutrophil count > or equal to 1500/ul, hemoglobin greater than or equal to 8.0 gm/dl, and platelets > than or equal to 100,000/ul.
* Adequate renal documented by serum creatinine < than or equal to 2.0 mg/dL
* Adequate hepatic function: Total serum bilirubin must be within institutional normal limits; transaminases (ALT and AST) may be up to 2.5 x institutional upper limit of normal (ULN) if alkaline phosphatase is < than or equal to ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are < than or equal to ULN.

If peripheral neuropathy is present, it must be less than or equal to grade 1

* Capable of providing written, informed consent
* Women with child-bearing potential must have a negative pregnancy test and must consent to using effective contraception while on treatment and for a reasonable period there after.

Exclusion Criteria:

* Active, or uncontrolled infection
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than 3 years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded. Patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than 3 years prior to registration, and that the patient remains free of recurrent or metastatic disease.
* With the exception of non-melanoma skin cancer and other specific malignancies as noted above, patients with other invasive malignancies who had (or have) any evidence of the other cancer present within the last 3 years or whose previous cancer treatment contraindicates this protocol therapy are excluded.
* Known history of hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80, or history of hypersensitivity reaction to gemcitabine.
* Currently has grade 2, 3 or 4 neuropathy
* Pregnant or lactating women
* Known history of congestive heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-08; Primary Completion 2006-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine the tolerability of delivering 4 cycles of docetaxel plus gemcitabine. | conclusion of the study

SECONDARY OUTCOMES:
Determine the percentage of pts with completely resected uterine LMS tx with the regimen that remain progression-free at 2 years, & compare this rate with historical controls to establish an estimate of the efficacy of the adjuvant treatment strategy. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Martee Hensley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org